CLINICAL TRIAL: NCT04415333
Title: Effect of Gut Butyrate Delivery on Blood Pressure in African Americans With Hypertension
Brief Title: Gut Butyrate and Blood Pressure in African Americans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other); North Carolina Agriculture & Technical State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 18-1680
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Hypertension
Keywords: African American; Blood pressure; Gut Microbiome; Short-chain fatty acid; Butyrate
MeSH Terms: conditions — Hypertension | interventions — Butyric Acid

STUDY DESIGN:
Intervention Model Description: In this blinded study, participants with Hypertension will self-administer a [5 mmol] and a [80 mmol] sodium butyrate enema in a randomized order 1 week (7 days) apart.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the participants with hypertension will perform the enema in a randomized order. The participants, nursing research staff (e.g., care providers), nor the PI's will know which enema the subjects are receiving. The study Biostatistician (e.g., statistical outcome assessor) will only be given the treatment IDs and not be given the sodium butyrate concentrations during statistical analyses. Randomization will be performed by 1 member of the research team at the beginning of the study who is also not involved in any informed consent process. Enemas will be assigned a letter (e.g., A or B) and each letter will be placed in an envelope (blinded allocation concealment). The research team member will reveal the key upon the conclusion of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sodium Butyrate [5 mmol] first, then Sodium Butyrate [80 mmol] (Experimental): After a randomized assignment in the crossover design, participants with hypertension will come to the testing office to self-administer the first enema with a concentration of 5 mmol sodium butyrate in a 0.9% saline solution (60 mL total). After a 7-days washout period, they will return to testing office to self-administer the other enema with a concentration of 80 mmol sodium butyrate in a 0.9% saline solution (60 mL total).
  Interventions: Drug: Sodium Butyrate 5 mmol; Drug: Sodium Butyrate 80 mmol
- Sodium Butyrate [80 mmol] first, then Sodium Butyrate [5 mmol] (Experimental): After a randomized assignment in the crossover design, participants with hypertension will come to the testing office to self-administer the first enema with a concentration of 80 mmol sodium butyrate in a 0.9% saline solution (60 mL total). After a 7-day washout period, they will return to the testing office to self-administer the other enema with a concentration of 5 mmol sodium butyrate in a 0.9% saline solution (60 mL total).
  Interventions: Drug: Sodium Butyrate 5 mmol; Drug: Sodium Butyrate 80 mmol
- Control (No Intervention): African Americans with normal blood pressure (control group) will not perform self-administration of the enema. They will submit to 1 blood draw and wear the 24-hour ambulatory blood pressure monitor for 1-day.

INTERVENTIONS:
Drug: Sodium Butyrate 5 mmol — Enema-based delivery of 5 mmol butyrate in 0.9% saline, (60 mL total)
  Arms: Sodium Butyrate [5 mmol] first, then Sodium Butyrate [80 mmol]; Sodium Butyrate [80 mmol] first, then Sodium Butyrate [5 mmol]
Drug: Sodium Butyrate 80 mmol — Enema-based delivery of 80 mmol butyrate in 0.9% saline, (60 mL total)
  Arms: Sodium Butyrate [5 mmol] first, then Sodium Butyrate [80 mmol]; Sodium Butyrate [80 mmol] first, then Sodium Butyrate [5 mmol]

SUMMARY:
African Americans have the greatest burden of hypertension. Recently, the short-chain fatty acid, butyrate, has been reported to have some effect on blood pressure. Butyrate is not normally ingested since it is made by bacteria in the gut as a byproduct of fiber fermentation. In this proof of concept study, the investigators will investigate the effect of butyrate absorbed in the gut (via the participant self-administering an enema with butyrate) has on blood pressure.

DETAILED DESCRIPTION:
Description: African Americans (AA) have the greatest burden of hypertension. Recently, gut microbial dysbiosis (a term that describes a poorly diverse gut microbial profile and lower short-chain fatty acid (SCFA) production) has been linked to hypertension and may be involved in the pathogenesis of hypertension in African Americans. African Americans have been reported to have lower gut SCFA and SCFA can reduce blood pressure. This is a proof of concept pilot study to determine the relationship between gut SCFA and blood pressure (BP). Delivery of butyrate to the gut will be via enema.

Objectives: The objectives of this research are to 1. Identify gut microbial taxa (SCFA butyrate-producing microbes) and circulating butyrate levels associated with hypertension via a cross-sectional design in AA without and with hypertension. 2. Quantify the relationship between SCFA (butyrate) absorption into the bloodstream and subsequent changes in blood pressure in a 24-hour period after delivering butyrate into the gut via enema.

Participants: African Americans males and females ages of 30-50 without hypertension (normal BP/healthy control; systolic BP: 90-129/ diastolic BP: 60-89mmHg) and with hypertension (systolic BP: 130-159 mmHg/ diastolic BP: 80-99 mmHg) that do not take anti-hypertension medication will be recruited.

Description of Study: There are 2 groups; control (without hypertension; BP: 90-129/60-89mmHg; 5 male/5 female, n=10) and experimental (with hypertension; BP 130-159/80-99 mmHg; 5 male/5 female, n=10). Normotensive participants (control group) will be age (±1 year) and sex-matched to hypertensive group participants. All participants (control and experimental groups; 5 male/5 female) will provide stool and blood samples, and complete 24-hour (hr) ambulatory blood pressure (ABP) monitoring to compare the abundance of fecal butyrate-producing microbes, circulating (blood) butyrate concentrations, and average blood pressure responses during the day and overnight. Individuals in the control group will only participate in donating stool (1-time) and a blood sample (1-time) and wearing a 24-hr ABP monitor (1-day). In a crossover blinded randomized controlled pilot study, the 10 hypertensive AA subjects (5 male/5 female) will be randomized to self-administer a sodium butyrate (80mmol butyrate in 0.9% saline, 60 ml total) or control (low dose) butyrate (5mmol butyrate 0.9%, 60 ml total) enema 1 week apart (7 days). Subjects will provide a stool sample before each study day (2 total), have their BP measured via ABP monitor, submit to a blood draws (pre-enema-baseline), self-administer the randomized enema, submit to a 30 min & 60 min post-enema blood draw, and wear the 24-hour ABP monitor for the remainder of that day. Subjects will be provided with written and verbal instructions on how to self-administer the enema. The dietary supplement (sodium butyrate) will be compounded by a local pharmacy (Custom Care Pharmacy - 109 Pisgah Church Rd. Greensboro, NC) into an enema at the concentrations listed above.

ELIGIBILITY:
Inclusion Criteria:

Normotensive (control subjects without hypertension): In order to be eligible to participate in this study, an individual must meet all of the following criteria (which will be assessed after an initial telephone interview and at Visit 1 (screening and consent visit):

* Provision of signed and dated informed consent form
* Be an African American adult (man or woman) between 30 - 50 years of age with normal blood pressure (never diagnosed with hypertension) (systolic: 90-129 and diastolic: 60-89 mmHg).
* Body Mass Index of 18.5-30 kg/m^2
* Not have any other diagnosed cardiovascular disease
* Not exercise regularly (Participate in less than 60 minutes of exercise/week)
* Not be pregnant or be lactating
* Be free of active diseases that affect your intestines (i.e., chronic constipation, diarrhea, Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, diabetes, hepatitis, HIV, and cancer)
* Have not taken antibiotics in the past 3 months
* Have not been regularly taking medications that impact intestinal function (i.e., laxatives, enemas, anti-diarrheal agents, narcotics, antacids, antispasmodics, antidepressants, anticonvulsants, antibiotics, herbals, homeopathy, and home remedies) or fiber supplements.
* Have no plans of travel out of town during the study periods.
* Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration

Hypertension subjects not on anti-hypertension medication (intervention group). The pool of subjects that do not take hypertension medication may be limited. If a heavily medicated subject population is encountered, the investigators may include subjects taking diuretics only: In order to be eligible to participate in this study, an individual must meet all of the following criteria (which will be assessed after an initial telephone interview and at Visit 1 (screening and consent visit):

* Provision of signed and dated informed consent form. Letter of clearance or signature of PCP on informed consent.
* Be an African American adult (man or woman) between 30 - 50 years of age with stage-1 to stage-2 hypertension (systolic: 130-159 and diastolic: 80-99 mmHg).
* Not taking any anti-hypertension medications (although the investigators may enroll individuals only taking a diuretic where resting BP levels are within the range of stage-1 hypertension: systolic BP 130-140 mmHg. Subjects can resume taking the diuretic after they remove the monitor).
* Body Mass Index of 18.5-30 kg/m^2
* Not have any other diagnosed cardiovascular disease
* Not exercise regularly (Participate in less than 60 minutes of exercise/week)
* Not be pregnant or be lactating
* Be free of active diseases that affect your intestines (i.e., chronic constipation, diarrhea, Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, diabetes, hepatitis, HIV, and cancer)
* Have not taken antibiotics in the past 3 months
* Have not been regularly taking medications that impact intestinal function (i.e., laxatives, enemas, anti-diarrheal agents, narcotics, antacids, antispasmodics, antidepressants, diuretics, anticonvulsants, antibiotics, herbals, homeopathy, and home remedies) or fiber supplements.
* Have no plans of travel out of town during the study periods.
* Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria for both groups:

* Exercise more than 60 minutes per week for more than 4 consecutive weeks.
* Diagnosed with stroke, history of myocardial infarction (heart attack); liver, lung, or kidney diseases; peripheral vascular disease or cancer within the last 6 months.
* Presence of metabolic disease (diabetes mellitus), inflammatory diseases (e.g., inflammatory bowel diseases, rheumatoid arthritis, and systemic lupus erythematosus); kidney stones or gallbladder problems; diagnosed liver, lung or kidney diseases;
* Pregnancy, lactation, or actively trying to conceive.
* Taking anti-hypertension medications (i.e., calcium channel blockers, ACE inhibitors, angiotensin- receptor blockers, β-blockers, vasodilators, etc.) other than diuretics (e.g., hydrochlorothiazide, chlorothiazide, furosemide, etc) or medications known to affect inflammation or metabolic function (anti-inflammatories, statins, thyroid medication) in the past 1 month. If diuretics are used, subjects may able to participate if they agree to refrain from taking their diuretic the day of the experiment. In this instance, resting systolic BP while on their medication will still need to be greater than 130 mmHg.
* Current smoker or tobacco use within the last 10 years

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc D Cook, PhD, Principal Investigator — North Carolina A&T State Univeristy
Locations (1):
- NC A&T State University, Greensboro, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share the informed consent and de-identified data set including fecal microbiome sequencing, blood pressure data, circulating butyrate levels in an online repository (Carolina Digital Repository).
Supporting Information: ICF
Time Frame: 3-5 years after the completion of the primary endpoint.
Access Criteria: Contact Dr. Marc Cook (mdcook@ncat.edu) at NC A&T State University. The data set will be shared in the Carolina Digital repository.
URL: https://library.unc.edu/scholarly-communications/open-access/carolina-digital-repository-cdr/

REFERENCES:
- [Background] Steinhart AH, Hiruki T, Brzezinski A, Baker JP. Treatment of left-sided ulcerative colitis with butyrate enemas: a controlled trial. Aliment Pharmacol Ther. 1996 Oct;10(5):729-36. doi: 10.1046/j.1365-2036.1996.d01-509.x. PMID 8899080
- [Background] Vanhoutvin SA, Troost FJ, Kilkens TO, Lindsey PJ, Hamer HM, Jonkers DM, Venema K, Brummer RJ. The effects of butyrate enemas on visceral perception in healthy volunteers. Neurogastroenterol Motil. 2009 Sep;21(9):952-e76. doi: 10.1111/j.1365-2982.2009.01324.x. Epub 2009 May 19. PMID 19460106
- [Background] Hamer HM, Jonkers DM, Vanhoutvin SA, Troost FJ, Rijkers G, de Bruine A, Bast A, Venema K, Brummer RJ. Effect of butyrate enemas on inflammation and antioxidant status in the colonic mucosa of patients with ulcerative colitis in remission. Clin Nutr. 2010 Dec;29(6):738-44. doi: 10.1016/j.clnu.2010.04.002. Epub 2010 May 15. PMID 20471725
- [Background] Krokowicz L, Stojcev Z, Kaczmarek BF, Kociemba W, Kaczmarek E, Walkowiak J, Krokowicz P, Drews M, Banasiewicz T. Microencapsulated sodium butyrate administered to patients with diverticulosis decreases incidence of diverticulitis--a prospective randomized study. Int J Colorectal Dis. 2014 Mar;29(3):387-93. doi: 10.1007/s00384-013-1807-5. Epub 2013 Dec 18. PMID 24343275
- [Derived] Hogue T, Das P, Reczek S, Hampton-Marcell J, Ford Y, Raval D, Carroll I, Cook MD. Effect of Acute Gut Butyrate Delivery on Blood Pressure in Black Individuals With Hypertension: A Proof-of-Concept Randomized Controlled Study. J Am Heart Assoc. 2025 Sep 2;14(17):e039759. doi: 10.1161/JAHA.124.039759. Epub 2025 Jul 30. PMID 40736085
- Available data/document: De-identified data set — https://library.unc.edu/scholarly-communications/open-access/carolina-digital-repository-cdr/ — Data will be accessible at the above Carolina Data Repository for the UNC library system.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sodium Butyrate [5 mmol] First, Then Sodium Butyrate [80 mmol]: After a randomized assignment in the crossover design, participants with hypertension will come to the testing office to self-administer the first enema with a concentration of 5 mmol sodium butyrate in a 0.9% saline solution (60 ml total). After a 7-day washout period, they will return to testing office to self-administer the other enema with a concentration of 80 mmol sodium butyrate in a 0.9% saline solution (60 ml total).
Period: First Intervention (Single 1-Day Visit)
Arm/Group | Sodium Butyrate [5 mmol] First, Then Sodium Butyrate [80 mmol] | Sodium Butyrate [80 mmol] First, Then Sodium Butyrate [5 mmol] | Control
Started (No participants received random assignment to the 80 mmol intervention first.) | 10 | 0 | 10
Completed | 10 | 0 | 10
Not Completed | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Sodium Butyrate [5 mmol] First, Then Sodium Butyrate [80 mmol] | Sodium Butyrate [80 mmol] First, Then Sodium Butyrate [5 mmol] | Control
Started | 10 | 0 | 10
Completed | 10 | 0 | 10
Not Completed | 0 | 0 | 0
Period: Second Intervention (Single 1-Day Visit)
Arm/Group | Sodium Butyrate [5 mmol] First, Then Sodium Butyrate [80 mmol] | Sodium Butyrate [80 mmol] First, Then Sodium Butyrate [5 mmol] | Control
Started | 10 | 0 | 10
Completed | 10 | 0 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants received random assignment to the 80 mmol intervention first.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sodium Butyrate [5 mmol] First, Then Sodium Butyrate [80 mmol] | Sodium Butyrate [80 mmol] First, Then Sodium Butyrate [5 mmol] | Control | Total
Number analyzed (Participants) | 10 | 0 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 0 | 10 | 20
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 6 | 11
  Male | 5 | 0 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 0 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 0 | 10 | 20
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 0 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Daytime Blood Pressure
Description: Immediately following self-administration of butyrate enema, participants will be fitted with an ambulatory blood pressure monitor to be worn for 24 hours.
Time Frame: approximately 16 hours post enema
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Sodium Butyrate [5 mmol]: Participants with hypertension self-administer an enema with a concentration of 5 mmol sodium butyrate in a 0.9% saline solution (60 mL total).
- Sodium Butyrate [80 mmol]: Participants with hypertension self-administer an enema with a concentration of 80 mmol sodium butyrate in a 0.9% saline solution (60 mL total).
Arm/Group | Sodium Butyrate [5 mmol] | Sodium Butyrate [80 mmol] | Control
Number analyzed (Participants) | 10 | 10 | 10
mmHg | 137.5 (13.47) | 132.9 (12.64) | 128.2 (16.31)

2. Primary Outcome: Mean Nighttime Blood Pressure
Description: as for outcome 1
Time Frame: approximately 8 hours post enema
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sodium Butyrate [5 mmol] | Sodium Butyrate [80 mmol] | Control
Number analyzed (Participants) | 10 | 10 | 10
mmHg | 123.2 (13.5) | 116.2 (10.9) | 114.0 (12.8)

3. Secondary Outcome: Blood Butyrate Concentrations
Description: Measure blood butyrate concentrations before, 30 minutes post, and 60 minutes post self-administration of the butyrate enemas
Time Frame: up to 1 hour post enema
Population: Unable to perform venipuncture for 1 participant in the control arm. Only baseline data are reported for the control arm for reference purposes as this group did not receive the intervention. Unable to collect blood at the 60-minute time point due to consistent antecubital vein rupturing after repeated venipuncture efforts.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sodium Butyrate [5 mmol] | Sodium Butyrate [80 mmol] | Control
Number analyzed (Participants) | 10 | 10 | 9
ng/mL
  Baseline | 143.88 (20.62) | 138.60 (16.84) | 149.89 (45.47)
  30 Minutes Post: number analyzed (Participants) | 10 | 10 | 0
  30 Minutes Post | 138.64 (11.29) | 151.57 (36.12) |
  60 Minutes Post: number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Interleukin-1 Beta (IL-1β) Concentration
Description: Blood biomarker samples were collected for the inflammatory cytokine IL-1β.
Time Frame: up to 1 hour post enema
Population: Insufficient sample collected to allow for analysis for 1 participant in the sodium butyrate (80 mmol) group and unable to perform venipuncture for 1 participant in the control arm.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sodium Butyrate [5 mmol] | Sodium Butyrate [80 mmol] | Control
Number analyzed (Participants) | 10 | 9 | 9
pg/mL | NA (NA) — IL-1β concentrations in every sample were below the detectable limit of 15.6 pg/mL | NA (NA) — IL-1β concentrations in every sample were below the detectable limit of 15.6 pg/mL | NA (NA) — IL-1β concentrations in every sample were below the detectable limit of 15.6 pg/mL

ADVERSE EVENTS:
Time Frame: During each 1-Day study visit through 24 hours post intervention administration and an additional 7 days after the final 1-Day study visit.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed for the control participants.
Groups:
- Sodium Butyrate (5 mmol): Participants with hypertension will come to the testing office to self-administer the first enema with a concentration of 5 mmol sodium butyrate in a 0.9% saline solution (60 ml total).
- Sodium Butyrate (80 mmol): Participants with hypertension will come to the testing office to self-administer the first enema with a concentration of 80 mmol sodium butyrate in a 0.9% saline solution (60 ml total).
Arm/Group | Sodium Butyrate (5 mmol) | Sodium Butyrate (80 mmol) | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/0
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/33/NCT04415333/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT04415333/ICF_000.pdf